CLINICAL TRIAL: NCT03177824
Title: Sildenafil Citrate for Treatment of Growth-restricted Fetuses
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohamed Ezz el din, resident of obstetrics and gynecology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 123sc
Record Dates: First submitted 2017-04-26; First posted 2017-06-06 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Fetal Growth Restriction
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- S (Experimental): Sildenafil citrate (25mg)
  Interventions: Drug: Sildenafil Citrate 25Mg Tab
- P (Placebo Comparator): placebo oral tablet
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Sildenafil Citrate 25Mg Tab — Group 1, consists of 30 patients who will receive Sildenafil citrate (25mg) tab (Silden, Epico, Egypt) 3times daily till the time of delivery, followed by repeating the Doppler US scan serially to detect changes in the measured indices and then assess the neonatal outcome after delivery as regard birth weight and APGAR score.
  Arms: S
Drug: Placebo Oral Tablet — Group 2, consists of 30 patients receiving placebo Oral Tablet 3times daily , followed by repeating the Doppler US scan serially to detect changes in the measured indices and then assess the neonatal outcome after delivery as regard birth weight and APGAR score
  Arms: P

SUMMARY:
The aim of this study is to assess the effect of Sildenafil citrate therapy on neonatal outcomes in women with fetal growth restriction.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age ranging from 20-40 years.
* Gestational age 28-37 weeks.

Exclusion Criteria:

* Obese patients (BMI >30 kg/m2).
* Patients with medical disorders: cardiac diseases, pulmonary diseases, liver disease, renal disease, previous history of seizures, hearing loss.
* Drug interactions, such as users of any vasodilator agents, omeprazole, clarithromycin and amoxicillin.
* Fetal distress.
* Pregnancy of multiple fetuses.
* Congenital fetal malformation or chromosomal abnormalities.
* Diastolic blood pressure more than 110 mmHg.
* Hypersensitivity to the drug.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-03-30 (Actual); Primary Completion 2017-09-30 (Estimated); Study Completion 2017-10-01 (Estimated)

PRIMARY OUTCOMES:
date of delivery after Sildenafil citrate administration. | for 6 months from the beginning of the study
  the study aims to assess date of delivery of growth restricted fetus after administration of sildenafil citrate by dose of 20mg three times per day , and that will be done by following up women with growth redistricted fetuses in Ain shams university maternity hospital till time of delivery.

SECONDARY OUTCOMES:
Expected fetal weight by serial ultrasound after Sildenafil citrate administration | every two weeks after drug intake for 6 months from the beginning of the study
  the Expected fetal weight in grams by serial ultrasound is assessed in women with growth redistricted fetuses in Ain shams university maternity hospital after Sildenafil citrate administration and till time of delivery .
Color Doppler changes on umbilical artery | weekly after drug intake for 6 months from the beginning of the study
  Color Doppler changes on umbilical artery is assessed in women with growth restricted fetuses in Ain shams university maternity hospital after Sildenafil citrate administration and till time of delivery .
neonatal outcomes as regard birth weight | for 6 months from the beginning of the study
  the study aims to assess neonatal outcomes as regard, birth weight in growth restricted fetus after administration of sildenafil citrate and that will be done by following up women with growth redistricted fetuses in Ain shams university maternity hospital till time of delivery.
neonatal outcomes as regard APGAR score | for 6 months from the beginning of the study
  the study aims to assess neonatal outcomes as regard APGAR score in growth restricted fetus after administration of sildenafil citrate and that will be done by following up women with growth redistricted fetuses in Ain shams university maternity hospital till time of delivery.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams matrnity hospital, Cairo, Egypt